CLINICAL TRIAL: NCT01955200
Title: Intensified Antiplatelet Therapy in Post-PCI Patients With High On-treatment Platelet Reactivity: the OPTIMA-2 Trial
Brief Title: OPTImal Management of Antithrombotic Agents: OPTIMA-2 Trial
Acronym: OPTIMA-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chunjian Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
Keywords: Stent implantation; High on-treatment platelet reactivity; Ticagrelor; Cilostazol; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Cilostazol; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CLOP-150 (Experimental): clopidogrel 150mg once daily
  Interventions: Drug: Clopidogrel
- CLOP+CILOST (Experimental): clopidogrel 75mg once daily plus cilostazol 100mg twice daily
  Interventions: Drug: Cilostazol
- TICAG (Experimental): ticagrelor 90mg twice daily
  Interventions: Drug: Ticagrelor
- CON(conventional DAPT) (Active Comparator): clopidogrel 75mg once daily
  Interventions: Drug: Clopidogrel
- Non-HOPR (Active Comparator): clopidogrel 75mg once daily
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — (ASA 100mg daily + Clopidogrel 150mg daily) x 1 month; (ASA 100mg daily + Clopidogrel 75mg daily) x 11 month.
  Other Names: Plavix
  Arms: CLOP-150
Drug: Cilostazol — (ASA 100mg daily + Clopidogrel 75mg daily + Cilostazol 150mg Bid) x 1 month; (ASA 100mg daily + Clopidogrel 75mg daily) x 11 month.
  Other Names: Peida
  Arms: CLOP+CILOST
Drug: Ticagrelor — (ASA 100mg daily + Ticagrelor 90mg Bid) x 1 month; (ASA 100mg daily + Clopidogrel 75mg daily) x 11 month.
  Other Names: Brilinta
  Arms: TICAG
Drug: Clopidogrel — (ASA 100mg daily + Clopidogrel 75mg daily) x 12 month.
  Other Names: Plavix
  Arms: CON(conventional DAPT)
Drug: Clopidogrel — (ASA 100mg daily + Clopidogrel 75mg daily) x 12 month.
  Other Names: Plavix
  Arms: Non-HOPR

SUMMARY:
High on-treatment platelet reactivity (HOPR) is associated with increased risk of cardiovascular events in patients undergoing percutaneous coronary intervention (PCI). We sought to investigate the efficacy and safety of 1-month intensified antiplatelet therapies in post-PCI patients with HOPR.

DETAILED DESCRIPTION:
OPTImal Management of Antithrombotic agents: OPTIMA-2 trial

Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor is the foundation antiplatelet therapy in patients undergoing percutaneous coronary intervention (PCI). Clopidogrel is the most commonly used P2Y12 receptor inhibitor worldwide because it is effective and inexpensive1. High on-treatment platelet reactivity (HOPR) occurs in as many as one-third of patients treated with standard dose clopidogrel (75mg once daily), and is associated with an increased risk of major adverse cardiovascular events (MACE).

Various approaches have been tested to overcome HOPR in patients treated with aspirin and clopidogrel, including higher doses of clopidogrel; the addition of cilostazol; and replacement of clopidogrel with prasugrel; however, the results of these intensified treatments were controversial, and a more potent P2Y12 receptor inhibitor, ticagrelor has never been studied in this scenario.

TOPIC study showed that short-term (i.e. 1-month) intensification of antiplatelet treatment might be sufficient to achieve optimal outcomes. Similarly, TROPICAL ACS showed that guided de-escalation of antiplatelet treatment with clopidogrel was non-inferior to the treatment with prasugrel at 1 year after PCI in terms of net clinical benefit, which suggests that routinely long-term intensification of antiplatelet treatment is not required for all PCI patients.

Accordingly we performed a randomized trial to test the hypothesis that in patients with HOPR intensification of antiplatelet therapy with double dose clopidogrel, the addition of cilostazol, or replacement of clopidogrel with ticagrelor for 1 month followed by resumption of conventional DAPT with aspirin and clopidogrel for 11 months would be superior to conventional DAPT for 12 months in reducing the prevalence of HOPR and MACE without increasing bleeding.

Inclusion criteria:

1. Successively recruit all patients who receive stent implantation;
2. Intended use of conventional DAPT with the combination of aspirin 100mg once daily and clopidogrel 75mg once daily for at least 12 months;
3. Patient aged over 18 years;
4. Signed inform consent.

Exclusion criteria:

1. Allergy or intolerance to study drugs;
2. History of gastrointestinal or intracranial bleeding;
3. Need for anticoagulant therapy;
4. High risk of bleeding (e.g., myelodysplasia, baseline platelet count < 80 × 109/L);
5. Hemoglobin < 90g/L;
6. Active malignancy or life expectancy < 1 year;
7. Patients with other conditions made them unsuitable to be recruited at the discretion of the investigators.

Study procedures:

Following treatment for at least 5 days with the combination of aspirin 100mg once daily and clopidogrel 75mg once daily irrespective of a loading dose we measured platelet aggregation in response to adenosine diphosphate (ADP) (PLADP) using light transmittance aggregometry (LTA). HOPR was defined as PLADP > 40%. Patients with HOPR were continued on aspirin 100mg once daily and were randomly assigned to one of the following 4 groups:

1. clopidogrel 150mg once daily (CLOP-150);
2. clopidogrel 75mg once daily plus cilostazol 100mg twice daily (CLOP+CILOST);
3. ticagrelor 90mg twice daily (TICAG);
4. clopidogrel 75mg once daily (conventional DAPT, CON). At 1 month, platelet aggregation testing was repeated after which all patients were switched back to conventional DAPT for a further 11 months.

All patients without HOPR were treated with conventional DAPT and followed to 12 months (Non-HOPR).

Sample size calculation:

Based on the published literature, we assumed a 38% rate of persistent HOPR in patients randomized to intensified treatment and 60% in those randomized to CON therapy. With a sample size of 81 per group, we calculated that we would have 80% power to detect this difference with a 2-sided P value of 0.05. After allowing for 20% study drug discontinuation rate at 1 month, we planned a sample size of 405 patients with HOPR.

Platelet Reactivity Assay

1. ADP-induced platelet aggregation: Light transmittancy aggregation (LTA) in response to 5μM ADP.
2. Blood sample collection time: baseline (more than 5 days after taking clopidogrel 75mg daily and aspirin 100mg daily), 1month after randomization.

Clinical follow-up:

Time points: 1month, 6month, and 1year after randomization.

The study endpoints:

The primary outcome was the proportion of patients with persistent HOPR at 1 month.

The secondary outcomes included a composite of MACE including cardiovascular death, nonfatal myocardial infarction (MI), ischemic stroke, target vessel revascularization (TVR), stent thrombosis (ST) and cardiac readmission during 12-month follow-up, and any bleeding defined by the Thrombolysis in Myocardial Infarction (TIMI) criteria.

ELIGIBILITY:
Inclusion criteria:

1. Successively recruit all patients who receive stent implantation;
2. Intended use of standard DAPT with the combination of aspirin 100mg once daily and clopidogrel 75mg once daily for at least 12 months;
3. Patient aged >18 years and ≦80 years old;
4. Signed inform consent.

Exclusion criteria:

1. Allergy or intolerance to study drugs;
2. History of gastrointestinal or intracranial bleeding;
3. Need for anticoagulant therapy;
4. High risk of bleeding (e.g., myelodysplasia, baseline platelet count < 80 × 109/L);
5. Hemoglobin < 90g/L;
6. Active malignancy or life expectancy < 1 year;
7. Patients with other conditions made them unsuitable to be recruited at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1724 (Actual)
Dates: Start 2013-10-05 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with persistent HOPR at 1 month | 1-month after randomization
  platelet aggregation in response to 5μM adenosine diphosphate (PLADP) measured by light transmittancy aggregometer (LTA) ; HOPR was defined as PLADP > 40%.

SECONDARY OUTCOMES:
MACE | 1-year after randomization
  a composite of MACE including cardiovascular death, nonfatal myocardial infarction (MI), ischemic stroke, target vessel revascularization (TVR), stent thrombosis (ST) and cardiac readmission during 12-month follow-up,revascularization, and stent thrombosis (ARC definition)

OTHER OUTCOMES:
Bleeding | 1-year after randomization
  any bleeding defined by the Thrombolysis in Myocardial Infarction (TIMI) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Main C, Palmer S, Griffin S, Jones L, Orton V, Sculpher M, Henderson R, Sudlow C, Hawkins N, Riemsma R. Clopidogrel used in combination with aspirin compared with aspirin alone in the treatment of non-ST-segment-elevation acute coronary syndromes: a systematic review and economic evaluation. Health Technol Assess. 2004 Oct;8(40):iii-iv, xv-xvi, 1-141. doi: 10.3310/hta8400. PMID 15461878
- [Background] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Background] Kronzon I, Feit F. Clopidogrel plus aspirin was effective but increased bleeding in acute coronary syndromes without ST-segment elevation. ACP J Club. 2002 Mar-Apr;136(2):45. No abstract available. PMID 11874270
- [Background] De Miguel A, Ibanez B, Badimon JJ. Clinical implications of clopidogrel resistance. Thromb Haemost. 2008 Aug;100(2):196-203. PMID 18690337
- [Background] Mehta SR, Tanguay JF, Eikelboom JW, Jolly SS, Joyner CD, Granger CB, Faxon DP, Rupprecht HJ, Budaj A, Avezum A, Widimsky P, Steg PG, Bassand JP, Montalescot G, Macaya C, Di Pasquale G, Niemela K, Ajani AE, White HD, Chrolavicius S, Gao P, Fox KA, Yusuf S; CURRENT-OASIS 7 trial investigators. Double-dose versus standard-dose clopidogrel and high-dose versus low-dose aspirin in individuals undergoing percutaneous coronary intervention for acute coronary syndromes (CURRENT-OASIS 7): a randomised factorial trial. Lancet. 2010 Oct 9;376(9748):1233-43. doi: 10.1016/S0140-6736(10)61088-4. PMID 20817281
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Background] Sibbing D, Aradi D, Jacobshagen C, Gross L, Trenk D, Geisler T, Orban M, Hadamitzky M, Merkely B, Kiss RG, Komocsi A, Dezsi CA, Holdt L, Felix SB, Parma R, Klopotowski M, Schwinger RHG, Rieber J, Huber K, Neumann FJ, Koltowski L, Mehilli J, Huczek Z, Massberg S; TROPICAL-ACS Investigators. Guided de-escalation of antiplatelet treatment in patients with acute coronary syndrome undergoing percutaneous coronary intervention (TROPICAL-ACS): a randomised, open-label, multicentre trial. Lancet. 2017 Oct 14;390(10104):1747-1757. doi: 10.1016/S0140-6736(17)32155-4. Epub 2017 Aug 28. PMID 28855078
- [Background] Deharo P, Quilici J, Camoin-Jau L, Johnson TW, Bassez C, Bonnet G, Fernandez M, Ibrahim M, Suchon P, Verdier V, Fourcade L, Morange PE, Bonnet JL, Alessi MC, Cuisset T. Benefit of Switching Dual Antiplatelet Therapy After Acute Coronary Syndrome According to On-Treatment Platelet Reactivity: The TOPIC-VASP Pre-Specified Analysis of the TOPIC Randomized Study. JACC Cardiovasc Interv. 2017 Dec 26;10(24):2560-2570. doi: 10.1016/j.jcin.2017.08.044. PMID 29268886
- [Derived] Ying L, Wang J, Li J, Teng J, Zhang X, Ullah I, Samee A, Xu K, Chen J, Xu L, Zhu H, Li J, Yang L, Wang F, Fan Y, Zhang J, Lu Y, Gong X, Shi L, Eikelboom JW, Li C. Intensified antiplatelet therapy in patients after percutaneous coronary intervention with high on-treatment platelet reactivity: the OPTImal Management of Antithrombotic Agents (OPTIMA)-2 Trial. Br J Haematol. 2022 Jan;196(2):424-432. doi: 10.1111/bjh.17847. Epub 2021 Oct 5. PMID 34611892
- [Derived] Wang J, Abdus S, Tan C, Gu Q, Yang M, Wang G, Shi L, Gong X, Li C. Serum uric acid level negatively correlated with the prevalence of clopidogrel low response in patients undergoing antiplatelet treatment with aspirin and clopidogrel. Nutr Metab Cardiovasc Dis. 2020 Nov 27;30(12):2215-2220. doi: 10.1016/j.numecd.2020.07.025. Epub 2020 Jul 24. PMID 32912788